CLINICAL TRIAL: NCT01004146
Title: A Study on the Preoperative Use of Incentive Spirometry in Morbidly Obese Patients Undergoing General Anesthesia
Brief Title: Pre-op Use of Incentive Spirometry in Obese Patients
Acronym: IS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Davide Cattano, Associate Proffessor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-08-0622
Record Dates: First submitted 2009-03-30; First posted 2009-10-29 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-12

CONDITIONS: Lung Function; Bariatric Surgery
Keywords: incentive spirometry; bariatric surgery; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): Patients assigned to the control group were educated on the proper technique of using the incentive spirometer and were instructed to use it for 3 breaths once per day to become able to use the device properly and consistently.
  Interventions: Procedure: Incentive Spirometry
- Experimental Group (Experimental): Patients assigned to the experimental group were instructed to use the spirometer by inhaling as slowly and deeply as possible in a set of 10 times and to repeat the process at least 5 times every day until the day of surgery.
  Interventions: Procedure: Incentive Spirometry

INTERVENTIONS:
Procedure: Incentive Spirometry — helps patient monitor their inspiratory tidal volume and assists in the preventing lower airway collapse

SUMMARY:
The purpose of this study is to evaluate the use of preoperative incentive spirometry (IS) as an aid to improve postoperative lung function. The hypothesis is that application of a standardized protocol of preoperative respiratory care teaching and exercise will improve lung performance that will subsequently result in prevention of postoperative pulmonary complications and that increasing the duration of preoperative use better improves lung mechanics postoperatively. The investigators propose to compare a patient population that uses IS as currently prescribed in the routine course of care (only to be familiar with preoperatively, but use postoperatively) against a population that uses IS with a standardized regimen for at least 3 days prior to the operation in terms of preoperative IS volumes, intraoperative pulmonary mechanics, postoperative IS volumes, and incidence of postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity
* bariatric surgery
* must be able to use incentive spirometer

Exclusion Criteria:

* BMI=<40 kg/m2
* current symptoms of obstructive sleep apnea or actively using continuous positive airway pressure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Cattano, M.D., Principal Investigator — University of Texas Medical School
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Patients assigned to the control group were educated on the proper technique of using the incentive spirometer to familiarize themselves with the device. Subjects were instructed to use it for 3 breaths once per day so that they would able to use the device properly and consistently. All patients in this group used the device at least 3 days prior to their surgical procedure.
- Experimental Group: Patients assigned to the experimental group were instructed to use the incentive spirometer by inhaling as slowly and deeply as possible in a set of 10 times and were asked to repeat the process at least 5 times every day until the day of surgery. All patients in this group used the device at least 3 days prior to their surgical procedure.
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 25 | 25
Have Incentive Spirometry Data | 21 | 20
Completed | 21 | 20
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (12.4) | 45.2 (12.3) | 45.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Incentive Spirometry Volume
Description: After the operation, the patients to be discharged on the same day were approached in the postanesthesia care unit (PACU) and requested to use the spirometer again. The volume (best out of 2 attempts) was recorded together with the same vital signs recorded preoperatively. Patients who were admitted to the hospital were requested to use the spirometer again on postoperative day 1. The largest IS volume (out of 2 attempts) was recorded. The data presented is the mean largest IS volume the day after surgery.
Time Frame: 1 week before surgery to the day after
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 21 | 20
cc | 1557.9 (814.67) | 1458.33 (613.87)

2. Secondary Outcome: Level of Compliance
Time Frame: 3 days to 2 weeks after clinic visit on the day of surgery
Reporting Status: Not Posted

3. Secondary Outcome: Oxygen Saturation
Time Frame: one week prior to surgery up to one day after
Reporting Status: Not Posted

4. Secondary Outcome: Heart Rate
Time Frame: one week prior to surgery to post operative day 1
Reporting Status: Not Posted

5. Secondary Outcome: Respiratory Rate
Time Frame: one week prior to surgery to post operative day 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control Group | Experimental Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

LIMITATIONS AND CAVEATS:
Our analysis was limited to measuring lung volumes up until postoperative day 1.Extending this study a few days postoperatively likely would allow us to achieve a better understanding of the course of respiratory function recovery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No